CLINICAL TRIAL: NCT06262581
Title: Neoadjuvant Tisleizumab(BGB-A317) for dMMR/MSI-H Non-late Stage Colorectal Cancer Patients
Brief Title: Neoadjuvant Tisleizumab(BGB-A317) for dMMR/MSI-H Non-late Stage CRC Patients Before Surgery
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Gong Chen, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-FXY-471
Record Dates: First submitted 2022-11-03; First posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: DMMR Colorectal Cancer; Anti PD-1; Immunotherapy
Keywords: CRC
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- dMMR/MSI-H stage I-III CRC patients (Experimental): Patients will accept 4 dose of Tisleizumab(BGB-A317) treatment after enrollment and the assessment of the therapeutic effect by clinicians would be finished after that. Once the patients has been qualified as cCR , they could be exempted for surgery and continued the watch and wait management. If the patient has been assessed as able to R0 surgery , then they would received surgery. Otherwise ,they would be excluded from the trial.
  Interventions: Drug: Tisleizumab(BGB-A317)

INTERVENTIONS:
Drug: Tisleizumab(BGB-A317) — 200mg i.v. q3w
  Other Names: surgery

SUMMARY:
According to the cancer statistics in 2020, colorectal cancer (CRC) remains a major public health issue worldwide, representing the third common cancer (10%) and second leading cause of death (9.4%) with 5-year survival rate approaching 65%. Meanwhile, 28.8% of the newly diagnosed cases and 30.3% of the CRC-related death occurs in China. Among all the CRC, stage I-III account for 75%. For the standard management for non-late stage(stage I-III) CRC patients, surgery including the primary site and local lymph nodes dissection has been the most important one. But for the high-risk stage II and locally-advanced stage III CRC, neoadjuvant or adjuvant therapy such as chemotherapy and radiotherapy plays a vital role in preventing the residual cancer cells to relapse and spread to distant sites after surgery. For the past decades, immunotherapy like anti-PD-1 and anti-CTLA4 checkpoint inhibitor achieves great process in solid tumor treatment especially for late-stage CRC. And Pembrolizumab and Nivolumab has been proved for dMMR/MSI-H late-stage-CRC by FDA. Combination of Ipilimumab and Nivolumab has achieved great success among the early-stage-CRC in NICHE study. The investigators here to carry out a phase II clinical trial to explore the safety and effect of single anti-PD-1 (Tisleizumab-BGB-A317 ) neoadjuvant treatment for non-late stage CRC patients.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide consents and agree to follow the trial requirement and assessment;
* Age >=18
* ECOG score: 0 or1
* Biopsy pathological diagnosis as MSI-H/dMMR( both IHC and PCR method required)
* Measurable and assessible primary tumor sites according to RECIST 1.1
* Able to provide 22ml peripheral blood for assessment for ctDNA
* With all organ function sufficient
* No bowel obstruction or fistula
* No previous chemotherapy, radiotherapy and immunotherapy accepted history
* Distant metastasis excluded before surgery by CT scan
* Contraception required for women for the whole enrollment time until 3 months after last dose of immunotherapy

Exclusion Criteria:

* self-autoimmune diseases history such as SLE
* People who using the immune suppressor
* Severe allergy to other mono-clone antibody
* Cerebral metastasis which hasn't be managed yet
* Hypertension(SBP>140mmHg，DBP>90mmHg)
* Uncontrolled diabetes(FBG>10mmol/L)
* Accepted anti-PD-1 or anti-PD-L1 immunotherapy in the past
* Uncontrolled heart diseases such as NYHA II heart failure, unstable angina , cardiac infarction in 1 year and arrhythmia
* Systemic inflammation which needs whole body treatment
* Urine routine: protein >=++ or 24hr urine protein>=1g
* Innate or acquired immune deficiency like HIV and HBV
* Enrolled in other clinical trial already
* Confirmed as metastasis before the surgery
* Other malignancies has been diagnosed before
* Tuberculosis
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-23 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
pathological complete regression rate | From enrollment to 1 year after surgery
  Patients without noninvasive or focal-invasive residues or involved lymph nodes should be considered as having achieved pCR. The rate is these patients over the whole group.

SECONDARY OUTCOMES:
CR rate | From enrollment to 1 year after surgery
  Patients with non-invasive or focal-invasive or involved lymph nodes which persists for 4 weeks after neoadjuvant immunotherapy. The rate of these patients over the whole group.
Major Pathological Response rate | From enrollment to 1 year after surgery
  Rate of the patients who had focal invasive and residue tumor site which less than 10% both in primary tumors and all lymph nodes.
Disease free survival | From enrollment to 1 year after surgery
  The time interval between the enrollment to the events such as relapse, distant metastasis and progressed occured.

CONTACTS AND LOCATIONS:
Overall Officials: Gong Chen, Prof, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided